CLINICAL TRIAL: NCT06358950
Title: A Phase 2, Parallel-Group, Dose-Range-Finding Study With Randomized Double-Blind Treatment and Open-Label Periods to Evaluate the Safety and Efficacy of ALKS 2680 in Subjects With Narcolepsy Type 1
Brief Title: A Study to Evaluate the Safety and Effectiveness of ALKS 2680 in Subjects With Narcolepsy Type 1 (ALKS 2680-201)
Acronym: Vibrance-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALKS 2860-201
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Narcolepsy Type 1
Keywords: Narcolepsy; Cataplexy; Orexin
MeSH Terms: conditions — Narcolepsy; Cataplexy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 4 mg ALKS 2680 (Experimental)
  Interventions: Drug: ALKS 2680
- 6 mg ALKS 2680 (Experimental)
  Interventions: Drug: ALKS 2680
- 8 mg ALKS 2680 (Experimental)
  Interventions: Drug: ALKS 2680
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 2680 — Oral tablet of ALKS 2680 for once daily administration
  Arms: 4 mg ALKS 2680; 6 mg ALKS 2680; 8 mg ALKS 2680
Drug: Placebo — Oral tablet containing matching placebo for once daily administration
  Arms: Placebo

SUMMARY:
The purpose of this research study is to assess the safety and efficacy of ALKS 2680 compared to placebo, including whether participants taking ALKS 2680 experience a greater decrease in sleepiness and a decrease in cataplexy ("sudden loss of muscle control"), compared to participants taking placebo alone.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Has a BMI ≥18 and ≤40 kg/m2
* Meets the diagnostic criteria of Narcolepsy type 1 according to ICSD-3-TR guidelines. Additionally, meets the following criteria:

  * Is HLA-DQB1*06:02-positive
  * Has residual excessive daytime sleepiness and cataplexy
* Is willing and able to discontinue any medications prescribed for the management of narcolepsy symptoms for at least 14 days and for the duration of study
* Is willing to adhere to additional protocol requirements

Exclusion Criteria:

* Significant comorbid medical conditions, including other sleep, cardiovascular, psychiatric, hepatic or other disorders may be exclusionary; eligibility will be determined on an individual basis by the study investigator
* Is currently pregnant, breastfeeding, or planning to become pregnant during the study
* Is currently enrolled in another clinical study (other than the parent study) or used any investigational drug or device within 30 days prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Mean Sleep Latency (MSL) on the Maintenance of Wakefulness Test (MWT) from baseline to Week 6 | Baseline to Week 6

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale (ESS) from baseline to Week 6 | Baseline to Week 6
  Epsworth Sleepiness Scale is a 4-point scale used to measure excessive sleepiness from 0 (would never doze) to 3 (high chance of "dozing)
Mean weekly cataplexy rate (WCR) as derived by subject cataplexy diary | Measured at Week 5 and 6
Incidence of adverse events | Up to 15 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Medical Director, MD, Study Director — Alkermes, Inc.
Locations (43):
- United States (28):
  - Alkermes Investigational Site, Los Angeles, California
  - Alkermes Investigational Site, Redwood City, California
  - Alkermes Investigator Site, San Francisco, California
  - Alkermes Investigational Site, Santa Ana, California
  - Alkermes Investigational Site, Aurora, Colorado
  - Alkermes Investigational Site, Colorado Springs, Colorado
  - Alkermes Investigational Site, Brandon, Florida
  - Alkermes Investigator Site, Brandon, Florida
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigator Site, Winter Park, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Macon, Georgia
  - Alkermes Investigational Site, Stockbridge, Georgia
  - Alkermes Investigator Site, Peoria, Illinois
  - Alkermes Investigator Site, Lansing, Michigan
  - Alkermes Investigator Site, Sterling Heights, Michigan
  - Alkermes Investigator Site, Lincoln, Nebraska
  - Alkermes Investigational Site, Middletown, New Jersey
  - Alkermes Investigational Site, Denver, North Carolina
  - Alkermes Investigational Site, Huntersville, North Carolina
  - Alkermes Investigator Site, Canton, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Dublin, Ohio
  - Alkermes Investigational Site, Wyomissing, Pennsylvania
  - Alkermes Investigational Site, Columbia, South Carolina
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, San Antonio, Texas
  - Alkermes Investigational Site, The Woodlands, Texas
- Australia (2):
  - Alkermes Investigator Site, Macquarie Park, New South Wales
  - Alkermes Investigator Site, Bedford Park, South Australia
- Belgium (3):
  - Alkermes Investigational Site, Alken
  - Alkermes Investigational Site, Bruges
  - Alkermes Investigational Site, Namur
- Alkermes Investigational Site, Prague, Czechia
- France (2):
  - Alkermes Investigational Site, Bordeaux
  - Alkermes Investigational Site, Montpellier
- Italy (3):
  - Alkermes Investigational Site, Bologna
  - Alkermes Investigational Site, Milan
  - Alkermes Investigational Site, Verona
- Netherlands (2):
  - Alkermes Investigational Site, Heemstede
  - Alkermes Investigational Site, Zwolle
- Spain (2):
  - Alkermes Investigational Site, Barcelona
  - Alkermes Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Vibrance-1 Study — https://vibrancestudies.com/?utm_source=ClinicalTrials&utm_medium=Referral&utm_content=Listing&utm_campaign=Listing_Vibrance1